CLINICAL TRIAL: NCT06687096
Title: The Effect of a Recipe Resource on Quality of Colonoscopy Bowel Preparation and Patient Experience
Brief Title: Effect of a Recipe Resource on Quality of Colonoscopy Bowel Preparation and Patient Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, selim demirci, Clinical physician, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: colonoscopydietbooklet
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2023-11

CONDITIONS: Bowel Preparation; Patient Experience; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: All elective colonoscopies were performed by two experienced endoscopists who were unaware of the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The booklet group (Experimental): The research protocol was explained during the colonoscopy appointment, and patients, when they agreed to follow their diet according to the recipe booklet, were accepted as part of the patient intervention group.
  Interventions: Other: A recipe booklet
- Control (Other): The control group consists of patients who prepared for colonoscopy with the standard low-residue diet list without being given a recipe booklet.
  Interventions: Other: standart diet list

INTERVENTIONS:
Other: A recipe booklet — A recipe resource with visuals in line with the low-residue diet recommendations given to patients before colonoscopy, including cooking instructions for the meals in the diet list.
  Arms: The booklet group
Other: standart diet list — patients prepared with a routine colonoscopy preparation scheme
  Arms: Control

SUMMARY:
This study aimed to provide a recipe resource with visuals in line with the low-residue diet recommendations given to patients before colonoscopy, including cooking instructions for the meals in the diet list. In this way, we aimed to minimize confusion regarding dietary restrictions during colonoscopy preparation and ensure full compliance with the diet list. Our hypothesis is that this approach may enhance compliance with current recommendations and improve the quality of bowel preparation.

DETAILED DESCRIPTION:
A total of 153 patients were included in this study. At the time of scheduling an outpatient colonoscopy, intervention group and control group were randomly assigned using a random-number generator for treatment allocation. The research protocol was explained during the colonoscopy appointment, and patients, when they agreed to follow their diet according to the recipe booklet, were accepted as part of the patient intervention group. A consent form was signed and collected. The nurse responsible for patient education in the endoscopy secretariat informed the patient that this booklet is an important component of bowel preparation and adhere strictly to the recipes in the booklet. The group who received the standard diet list and applied for their colonoscopy appointments were randomly designated as the control group. Bowel preparation was evaluated during the colonoscopy using the Boston Bowel Preparation Scale (BBPS). Cecal insertion and withdrawal times, polyp detection rate, utilization of the recipe resource, and patients' experiences related to colonoscopy were recorded.

The research team utilized freely available resources from general cookery recipe websites to create the recipe resource, adapting it to align with the recommendations for a low-residue diet (figure). Recipes were selected based on criteria such as being visually appealing, easy to prepare, and easily modifiable to comply with the low-residue diet. A dietitian examined the recipe resource to guarantee that the recipes followed low-residue diet guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All outpatients who apply for a colonoscopy appointment.

Exclusion Criteria:

* Patients with a history of prior colonoscopic procedures
* Using anticholinergic or gastrointestinal motility-reducing drugs
* Severe chronic kidney failure (GFR<30 ml/min)
* Advanced heart failure (NYHA III-IV)
* History of abdominal surgery were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale (BBPS) | immediately after the procedure
  The BBPS is used to evaluate the quality of bowel preparation, with a scale from 0 to 9 (0 = very poor, 9 = excellent). Total BBPS score ≥ 6 and three segments of the colon (right, transverse, and the left side of the colon) ≥ 2 accepted as good bowel preparation

SECONDARY OUTCOMES:
patient experience | immediately after the procedure
  The patient experience of the study group was evaluated using a 3-point scale (1-worse than expected, 2-as expected, 3-better than expected).

CONTACTS AND LOCATIONS:
Overall Officials: selim demirci, medical doctor, Principal Investigator — Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Locations (1):
- Abdurrahman Yurtaslan Oncology and Training Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tae JW, Lee JC, Hong SJ, Han JP, Lee YH, Chung JH, Yoon HG, Ko BM, Cho JY, Lee JS, Lee MS. Impact of patient education with cartoon visual aids on the quality of bowel preparation for colonoscopy. Gastrointest Endosc. 2012 Oct;76(4):804-11. doi: 10.1016/j.gie.2012.05.026. Epub 2012 Jul 27. PMID 22840295
- [Background] Spiegel BM, Talley J, Shekelle P, Agarwal N, Snyder B, Bolus R, Kurzbard N, Chan M, Ho A, Kaneshiro M, Cordasco K, Cohen H. Development and validation of a novel patient educational booklet to enhance colonoscopy preparation. Am J Gastroenterol. 2011 May;106(5):875-83. doi: 10.1038/ajg.2011.75. Epub 2011 Apr 12. PMID 21483463
- [Background] Bennett L, Knox R, Luscombe G, Egan J, Wallace L. The Colonoscopy Cookbook: Analysis of effect of a recipe resource on quality and experience of bowel preparation in colonoscopy. Endosc Int Open. 2023 May 26;11(5):E561-E565. doi: 10.1055/a-2057-4374. eCollection 2023 May. PMID 37251792